CLINICAL TRIAL: NCT03586063
Title: A Multicenter Observational Study of Diphereline 3.75 mg Treatment Effectiveness in Russian Women Suffering From Internal Genital Endometriosis
Brief Title: Study of Diphereline 3.75 mg Treatment In Women Suffering From Internal Genital Endometriosis
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52014-191
Record Dates: First submitted 2018-06-08; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Internal Endometriosis
MeSH Terms: conditions — Adenomyosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — This is a non-interventional (observational) national multicentre prospective study.
  Treatment was administered according to the Summary of Product Characteristics (SmPC): maximum 6 injections administered every 28 days.
  The decision to prescribe GnRH-a (Diphereline 3,75 mg) was made prior to and independently from the decision to enroll the patient into the study.

SUMMARY:
To describe Gonadotropin-Releasing Hormone agonists (GnRH-a) treatment effectiveness on reduction of internal genital endometriosis symptom - menorrhagia - in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3,75 mg - assessment performed six months after the last injection.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 25-40 years old
* With symptomatic internal genital endometriosis - at least mild menorrhagia present or worse
* Internal genital endometriosis diagnosis is based on enlarged uterus detected by pelvic bimanual examination and ultrasound examination (stages I-II-III by Demidov in accordance with ultrasound results not earlier than 2 months before first injection
* Naive patients who have never been prescribed a GnRH agonist

Exclusion Criteria:

* Pregnant subjects
* Subjects with hypersensitivity to GnRH analogue or to one of its excipients
* Subjects treated with any other investigational drug within the last 30 days before study entry
* Subjects' refusal to participate in the study

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Antenatal clinics and Medical centres
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2011-11-03 (Actual); Primary Completion 2014-12-24 (Actual); Study Completion 2014-12-24 (Actual)

PRIMARY OUTCOMES:
Severity of disease symptom menorrhagia (none-mild-moderate-severe) in different disease stages I, II, III in the Russian subject population scheduled for treatment with Diphereline 3.75 mg | Change from baseline to up to 6 months after the last injection (up to month 11)
  A responder is defined as a subject with menorrhagia reduction at least by one level (i.e. from severe to moderate, from moderate to mild, from mild to none).

SECONDARY OUTCOMES:
Patients' age at study entry | Baseline (Day 1)
Age at the time of internal genital endometriosis diagnosis | Baseline (Day 1)
Gynaecological history | Baseline (Day 1)
  Age of menarche, hereditary load in onco-gynaecology, sexually transmitted infections, gynaecological surgical procedures, number of pregnancies, medical abortions, miscarriages, normal deliveries, coexisting gynaecological diseases, somatic diseases, if any.
Data on fertility: primary and secondary sterility | Baseline (Day 1)
Medical history | Baseline (Day 1)
Concomitant medications and non drug therapy for internal endometriosis treatment | Baseline (Day 1)
Severity of disease symptom dysmenorrhea (none-mild-moderate-severe) in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3.75 mg | On the day of the last injection (up to Month 5)
  A full responder is defined as the person with a reduction of intensity of at least one level for all symptoms of at least mild intensity at baseline (i.e. from severe to moderate, from moderate to mild, from mild to none).
Severity of disease symptom menorrhagia (none-mild-moderate-severe) in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3.75 mg | On the day of the last injection (up to Month 5)
  A full responder is defined as the person with a reduction of intensity of at least one level for all symptoms of at least mild intensity at baseline (i.e. from severe to moderate, from moderate to mild, from mild to none).
Severity of disease symptom metrorrhagia (none-mild-moderate-severe) | On the day of the last injection (up to Month 5)
  A full responder is defined as the person with a reduction of intensity of at least one level for all symptoms of at least mild intensity at baseline (i.e. from severe to moderate, from moderate to mild, from mild to none).
Severity of disease symptom pelvic pain (none-mild-moderate-severe) in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3.75 mg | On the day of the last injection (up to Month 5)
  A full responder is defined as the person with a reduction of intensity of at least one level for all symptoms of at least mild intensity at baseline (i.e. from severe to moderate, from moderate to mild, from mild to none).
Uterine volume in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3.75 mg | Baseline (Day 1) and on the day of the last injection (up to Month 5)
  Measured by ultrasound and calculated by the equation 0,523 x a x b x c, where a, b and c stand for uterine length, width and thickness, respectively
Uterine shape (bimanual pelvic examination) in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3.75 mg | Baseline (Day 1) and on the day of the last injection (up to Month 5)
Internal genital endometriosis symptom metrorrhagia in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3.75 mg | Change from baseline (Day 1) to 6 months after the last injection (up to Month 11)
Internal genital endometriosis symptom dysmenorrhea in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3.75 mg | Change from baseline (Day 1) to 6 months after the last injection (up to Month 11)
Internal genital endometriosis symptom pelvic pain in different disease stages I, II, III in the Russian patient population scheduled for treatment with Diphereline 3.75 mg | Change from baseline (Day 1) to 6 months after the last injection (up to Month 11)
Reproduction function will be assessed by the number of patients got pregnant 6 and 9 months after the end of treatment with Diphereline 3.75mg | 6 and 9 months after the end of treatment with Diphereline
Reproduction function will be assessed by the number of patients who avoided hysterectomy/ did not receive a surgical treatment 6 and 9 months after the end of treatment with Diphereline 3.75mg | 6 and 9 months after the end of treatment with Diphereline
Diphereline 3.75 mg treatment practice will be assessed by the number of scheduled/ performed injections with treatment schedule (each 28 days) in line with treatment administration approved in Russian Federation | Up to Month 5
Diphereline 3.75 mg treatment practice will be assessed by patient compliance with treatment schedule (each 28 days) in line with treatment administration approved in Russian Federation | Up to Month 5

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (34):
- Russia (34):
  - Moscow regional perinatal center, Balashikha
  - Scientific center of Family Health Problems and Human reproduction of Siberian branch of RAMS, Irkutsk
  - SEI Irkutsk State medical refresher institute, Irkutsk
  - Municipal healthcare institution "City hospital #11", Kazan'
  - City hospital #2, Krasnodar multi-field medical diagnostic association, endoscopic gynecology center, Krasnodar
  - SHI "Regional clinical hospital #1 named after S. Ochapovskiy", Krasnodar
  - SHI "City Clinical Hospital #79", Moscow
  - FSBI "Research Center of Obstetrics, Gynecology and Perinatology named after V. Kulakov" on the base of City clinical hospital named after S. Botkin, Moscow
  - Treatment rehabilitation Center of Roszdrav, Moscow
  - Central Clinical Hospital of Civil aviation, Moscow
  - CM-Clinic, Moscow
  - SI "Endocrinology Research Center" of the Ministry of Health and Social Development of the Russian Federation, Moscow
  - FBHI "Volga regional medical center" of Federal Medical-Biological agency, gynecological department of clinical hospital #1, Nizhny Novgorod
  - Non-governmental healthcare institution "Road clinical hospital on Gor'kiy station RZhD NChS, Nizhny Novgorod
  - Center of new medical technologies in academic town, Novosibirsk
  - Medical Center Zdravitsa, Novosibirsk
  - Fertility Clinic, Novosibirsk
  - Clinical hospital №123 of FMBA of Russia, Odintsovo
  - SHI "City hospital #8", Rostov-on-Don
  - Clinical hospital #1 of FSI "Southern federal district medical center", Rostov-on-Don
  - Rostov state medical university, department of obstetrics and gynaecology #3, based on SHI "Region hospital #2", Rostov-on-Don
  - SHI "Regional hospital #2", Rostov-on-Don
  - FSI "Rostov Research institution of obstetrics and pediatry", Rostov-on-Don
  - City hospital #3 of the Holy Reverend Martyr Elizabeth, Saint Petersburg
  - North-West State Medical University named after I. Mechnikov on the base of maternity hospital #17, Saint Petersburg
  - Scientific-Research Institute of obstetrics and gynecology named after D.O. Otto of Russian Academy of Medical Science, Saint Petersburg
  - Medical centre IDK, Samara
  - Non-governmental healthcare institution " Railway Clinical Hospital", Saratov
  - SHI "Regional Clinical Hospital", Saratov
  - SHI Saratov Regional Centre of Family Planning and Reproduction, Saratov
  - Non-governmental healthcare institution "Departmental clinical hospital on station Ufa RZHD", Ufa
  - Federal State-Funded Educational Institution of Higher Vocational Education "Volgogradskii State Medical University of Roszdrav on the base of Hospital #1, Volgograd
  - Medical center "Yunona", Yaroslavl
  - Municipal clinical healthcare Institution of Yaroslavl region "Primary healthcare unit NYa ORP", Yaroslavl